CLINICAL TRIAL: NCT03918785
Title: Rice Germ Supplementation on Moderately Trained Swimmers: a Randomized Pilot Clinical Trial
Brief Title: Rice Germ Supplementation on Swimmers
Acronym: RGS swimmers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Principal Investigator, Mariangela Rondanelli, Principal Investigator, Azienda di Servizi alla Persona di Pavia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1114/06072014
Record Dates: First submitted 2019-03-27; First posted 2019-04-18 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Athletes; Sports
Keywords: rice germ; swimmers; nutritional supplement; lactic acid; fat free mass

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rice Germ (Experimental): The Rice Germ was supplied in vacuum jars of a weight of 130 grams. These jars once opened, were stored in the refrigerator (-3-4°C). Together with cans, small containers were provided to act as dosers and served to determine the correct dose to be taken (25 grams, twice a day). The rice germ or placebo were continually taken every day twice a day (25 grams in the morning with breakfast and 25 grams in the afternoon as snacks) for 5 weeks. The rice germ was supplied by the company "Acquerello" (TenutaColombara, Livorno Ferraris, Vercelli, Italy).
  Interventions: Dietary Supplement: Rice germ
- Control group (Active Comparator): Active comparator, which consisted of an isocaloric wheat germ-based supplement. Characteristics of supplementation are the same of experimental group.
  Interventions: Dietary Supplement: Wheat-based supplement

INTERVENTIONS:
Dietary Supplement: Rice germ — 25 g twice a day.
  Arms: Rice Germ
Dietary Supplement: Wheat-based supplement — 25g twice a day.
  Arms: Control group

SUMMARY:
In order to enhance the effects of training and improve performance, athletes often turn to nutritional supplements. According to the American College of Sports Medicine (ACSM), adequate selection of nutrients and supplements, adjusting intake according to the exercise performed, is necessary for optimal performance in athletes. The most recent consensus from the International Society for Sport Nutrition (ISSN), The American Dietetic Association (ADA) and ACSM on sport nutrition have been reviewed by Potgieter, stating that a single guideline is not sufficient to elaborate an individualized and focused nutritional management of athletes. Moreover, apart from the abovementioned guidelines, sport-specific nutritional strategies, including quantity, structure and timing of food (or supplement) intake should also be followed in order to maximize sports performance and recovery. The importance of dietary supplementation is of particular interest in swimming, where athletes usually undertake a training approach characterized by a high volume of training during aerobic development and high intensity training during the competition phase, coupled with strength training.

The size and market value of the sports supplement industry is continuing to grow, with health, safety and contamination concerns becoming more pressing. Therefore, it is important to identify dietary supplements that are safe and effective in supporting swimmers. Rice germ could be a safe and effective dietary supplement for swimmers. In the last few years, scientific research is trying to use waste rice products in the pharmaceutical and nutraceutical fields, considering the potential value of nutrients they contain. In particular, rice germ has a high protein and essential amino acids, such as lysine, histidine and valine content, a good lipid content (with prevalence of mono- unsaturated and polyunsaturated fatty acids - in particular linoleic and linolenic essential fatty acids and oleic acid), an high fiber presence; regarding water-soluble vitamins, rice germ has high content if thiamine (B1) and pyridoxine (B6), while vitamin E prevails for liposoluble vitamins. About minerals, are most present iron and magnesium. All these nutrients play important roles in maintaining the health of athletes. Currently, despite these characteristics, no study has evaluated the potential beneficial effect of RG supplementation on athletes. Given this background, the purpose of this investigation was to ascertain whether performance in swimmers could be improved by a 5-weeks of RG supplementation.

ELIGIBILITY:
Inclusion Criteria:

* moderately trained athletes
* regularly involved in regional and national competitions

Exclusion Criteria:

* No history of cardiac or respiratory disease
* no medication at the time of the study
* no abnormalities on physical examination or on resting electrocardiogram

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Performance change | At baseline and after 5 weeks of supplementation
  Whether the performance in 50m, 200m, is improved in a 25m swimming pool in front crawl at maximal speed. Performance measured in seconds.
Lactic acid production change | At baseline and after 5 weeks
  Capillary blood samples were collected from the fingertip before and after each swimming (at the 1st and 3rdmin of recovery) to access the higher values of blood lactate concentration (AccutrendLactate®Roche, Germany).

SECONDARY OUTCOMES:
Antropometric measures change (skinfolds) | At baseline and after 5 weeks of supplementation
  skinfolds thicknesses (mm) (biceps, triceps, suprailiac, subscapular), measured twice using a Harpenden skinfold caliper at 5 min intervals at each site
Body weight change (kg) | At baseline and after 5 weeks of supplementation
  Change in body weight (kg).
Antropometric measures change (circumferences) | At baseline and after 5 weeks of supplementation
  Waist circumference (cm), hip circumference (cm), mid-arm circumference (cm).
Change in Total fat mass, total free fat mass and visceral adipose tissue (DXA) | At baseline and after 5-weeks of supplementation
  Body composition by dual-energy X-ray absorptiometry (DXA). Body composition was measured at baseline by DXA, using a Lunar Prodigy DEXA (GE Medical Systems, Waukesha, WI). Free Fat mass, Fat mass and visceral fat (kg) data were derived from DXA using the DXA Prodigy enCORE software (version 17; GE Healthcare).
Body composition parameters change (BIVA) | At baseline and after 5-weeks of supplementation
  Body composition analyzed with BIVA: free fat mass, fat mass, body cellular mass change (kg).
Hydration parameters change (BIVA) | At baseline and after 5-weeks of supplementation
  Hydration analyzed with BIVA: total body water, extracellular water, intracellular water change (L)
Registration of adverse effects | After 7 days, 14 days, 21 days, 28 days from baseline and after 5 weeks.
  Adverse effects recorded, through phone call
Muscle function change | At baseine and after 5 weeks.
  The JAMAR Hand Dynamometer (Jamar 5030J1; Sammons Preston Rolyan; accuracy 0.6 N) was used to assess muscle function with the use of a standardized procedure(Spijkerman, Dorine C., Snijders, Chris J., Stijnen, Theo, & Lankhorst 1991). Handgrip measured in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Rondanelli, MD, PhD, Professor, Study Director — Mariangela Rondanelli, IRCCS Mondino Foundation, Pavia

IPD SHARING:
Plan to Share IPD: No